CLINICAL TRIAL: NCT03367442
Title: Driving Pressure in Trauma. Morbi-mortality and Pulmonary Mechanics in Relation to Transpulmonary Driving Pressures in Patients With Chest Trauma. A Prospective Observational Study
Brief Title: Driving Pressure in Trauma
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0354
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Sever Chest Trauma; Mechanical Ventilation
Keywords: Thoracic trauma; mechanical ventilation; Acute respiratory distress syndrome; Esophageal pressure; Pleural pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Traumatic chest injuries are responsible for significant morbidity and the cause of trauma-related death in 20%-25% of cases. Thoracic trauma can include multiple injuries, mainly osseous (ribs, sternal fractures, flail chest), pulmonary contusions or lacerations, pneumothoraces and pleural effusions, and sometimes involve wounds to the heart and vessels (aortic dissection, cardiac contusion) or diaphragm. Following trauma, patients with thoracic injuries are at risk of developing acute respiratory distress syndrome (ARDS). This worsening of respiratory function can lead to requirement for mechanical ventilation. In addition, changes to gas exchange may also be generated or aggravated by mechanical ventilation as a result of barotrauma, biotrauma, or ventilation-associated pneumonia. Many mechanical ventilation strategies have been tried in trauma patients in the last 30 years to determine the optimal method of maximizing gas exchange with minimal lung damage. The driving pressure of the respiratory system has been shown to strongly correlate with mortality in a recent large retrospective ARDSnet study. Respiratory system driving pressure [plateau pressure-positive end-expiratory pressure (PEEP)] does not account for variable chest wall compliance especially in cases of chest trauma. Esophageal manometry can be utilized to determine transpulmonary driving pressure. A recent study suggests that utilizing PEEP titration to target positive transpulmonary pressure via esophageal manometry causes both improved elastance and driving pressures. Treatment strategies leading to decreased respiratory system and transpulmonary driving pressure at 24 h may be associated with improved 28 day mortality. However, currently no specific study with chest trauma patients exists. We propose to investigate the effect of hight transpulmonary driving pressure on duration on mechanical ventilation, length of stay and mortality in patients with sever chest trauma.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (18-90 years old)
* Affiliated to the social security
* Hospitalized following severe trauma chest trauma
* Mechanical ventilatory support for a minimum of 72 hours

Exclusion criteria:

* Minor patients,
* Patients under tutorship / curatorship,
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sever chest trauma under mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical Ventilation | 1 day
  Duration of mechanical Ventilation

SECONDARY OUTCOMES:
During of SDRA | 1 day
  During of SDRA
Length of stay in intensive care unit | 1 day
  Length of stay in intensive care unit
Mortality | 1 day
  Mortality
Pulmonary compliance | 1 day
  Pulmonary compliance
Pulmonary stress and strain | 1 day
  Pulmonary stress and strain

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan CHARBIT, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC